CLINICAL TRIAL: NCT06687421
Title: Swedish Prostate Cancer Initiative for Novel Treatment Regimens - Real, Implementation of Precision Medicine in High-risk Prostate Cancer
Brief Title: Implementation of Precision Medicine in High-risk Prostate Cancer
Acronym: SPRINTR-REAL
Status: Recruiting | Type: Observational
Sponsor: Andreas Josefsson (Other Government)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor-Investigator, Andreas Josefsson, Associate Professor / Urologist, Region Västerbotten
Organization: Region Västerbotten (Other Government)
Other Study IDs: SPRINTR-REAL
Record Dates: First submitted 2024-10-16; First posted 2024-11-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Androgen Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue from diagnostic prostate biopsies for whole genome RNA and DNA sequencing and tissue evaluations (immunohistochemistry, digital pathology). In selected groups (primarily non-metastatic high risk PC) blood and urine will be sampled for analysis/identification of biomarkers as liquid biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Non-metastatic high-risk prostate cancer: ISUP ≥4, T3-4, or regional lymph node positive
  Interventions: Other: High-risk treatment SOC
- Low risk prostate cancer: ISUP = 1, PSA <10 µg/L, PSA-density <0,15 µg/l/cm3
  Interventions: Other: Active monitoring
- Medium risk prostate cancer: ISUP 2-3, PSA 10-20 µg/L
  Interventions: Procedure: Radical prostatectomy; Radiation: Radiotherapy
- Metastatic prostate cancer: PSA > 80 µg/L, clinically manifest metastases
  Interventions: Drug: Androgen deprivation therapy

INTERVENTIONS:
Other: High-risk treatment SOC — radiotherapy (RT) + ADT (3 years) + Abiraterone acetate (2 years), with radical prostatectomy being an option if contraindication for RT exists)
  Groups: Non-metastatic high-risk prostate cancer
Other: Active monitoring — Followed with PSA measurements
  Groups: Low risk prostate cancer
Procedure: Radical prostatectomy — Radical prostatectomy
  Groups: Medium risk prostate cancer
Radiation: Radiotherapy — Radiotherapy
  Groups: Medium risk prostate cancer
Drug: Androgen deprivation therapy — GnRH agonist + abiraterone acetate/enzalutamide and/or docetaxel
  Groups: Metastatic prostate cancer

SUMMARY:
This project's objective is to initiate a prospective non-interventional clinical study to perform full molecular characterization and subtyping of the primary tumor prostate cancer patients.

It will identify, compare, and select biomarkers for treatment response in high-risk/metastatic prostate cancer.

DETAILED DESCRIPTION:
This prospective study includes molecular characterization of the primary tumor, biobanking of urine and blood, questionnaires, collection of health economic parameters, cross-checking of registries to link both other diagnoses and drug use to the different biomarkers and socio-economic parameters.

Clinical variables including imaging and routine pathology and the outcome of the molecular diagnostic analysis should, in addition to the basic scientific purpose, also be able to identify men who may be eligible for other studies, both pharmaceutical company-funded and investigator-initiated studies.

One aim is also to develop the national medical information system already in place for prostate cancer (individual patient record) with molecular profiling and other variables for health estimation, health economics and also enable retrieval from more registries.

This study will form the basis for the start of a nationwide study with the aim to prioritize biomarkers for the development of treatment predictive algorithms

ELIGIBILITY:
Inclusion Criteria:

* Men investigated for suspected prostate cancer
* Signed consent form

Exclusion Criteria:

* Difficulties understanding information about the study due to linguistic, cognitive or other reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All men who come for biopsy as a part of the investigation for suspected prostate cancer will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2054-12 (Estimated); Study Completion 2054-12 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | From enrollment to 20 years failure-free survival

SECONDARY OUTCOMES:
Biomarker profiling | From enrollment to 20 years.
  Molecular and imagebased characterization of primary tumor. RNA-sequencing, DNA -sequencing, whole genome arrays, analysis of immunohistochemical markers such as Ki67, PSA and AR will be performed as well as MR and PSMA-PET imaging.
EORTC QLQ-C15-PAL | From enrollment to 20 years.
  Questionnaire on quality of life
IPSS | From enrollment to 20 years
  Questionnaire on symptoms related to the prostate
Costs for implementing precision medicine | Before and after implementation of precision medicine workflows
  Evaluation of costs for implementing precision medicine tools including tumor profiling in the clinical workflow. Registration of all time required for handling of patient samples from referral to the clinic until diagnosis decision and cost for preparation/analysis of tissue for molecular characterization.
Cost effectiveness analysis | From enrollment to 20 years
  Evaluation of health economical costs measured by both crude costs for precision medicine workflow plus specific targeted treatments with or without quality-adjusted life years analysis. Data will be collected from health registries and surveys for quality of life evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology, Umeå University Hospital, Region Västerbotten, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All collected research data apart from identifiable data can be shared pseudonymised.
  In most cases results will be presented at group level. However if analysis results at the individual level will be presented baseline information will be presented in the form of intervals to prevent the research subject from being identified. Baseline information could be e.g. age and lab values. Therefore shared data will not be directly traceable to an individual participant.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting Jan 2025. Unending.
Access Criteria: Proposal that describes planned analyses must be submitted and a data sharing agreement must be signed.